CLINICAL TRIAL: NCT03401398
Title: Stress Hydrocortisone In Pediatric Septic Shock
Acronym: SHIPSS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jerry Zimmerman (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Critical Care Trials Group (Other); Children's Hospital of Eastern Ontario (Other)
Responsible Party: Sponsor-Investigator, Jerry Zimmerman, Professor of Pediatrics/Anesthesiology, University of Washington School of Medicine, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-P00027662; 1R01HD096901-01 (NIH)
Record Dates: First submitted 2018-01-05; First posted 2018-01-17 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-05

CONDITIONS: Septic Shock
Keywords: hydrocortisone; refractory septic shock; sepsis; new/progressive MODS; mortality; health-related quality of life; corticosteroid adverse events; sepsis biomarkers
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Hydrocortisone; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients randomized to the hydrocortisone treatment arm will receive an initial bolus of 2 mg/kg IV hydrocortisone (maximum 100 mg), followed by 1 mg/kg (maximum 50 mg) of hydrocortisone dosed every six hours for a maximum of seven days or until all vasoactive infusions have been discontinued for at least 12 hours, whichever comes first. When the hydrocortisone course is completed, the medication will be discontinued. Patients randomized to the placebo treatment arm will receive an equivalent volume of normal saline, with the identical dosing schedule outlined above.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects, families, critical care providers and investigators will be blinded to study drug administration. Only the local performance site research pharmacist will be un-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Approximately half of the subjects randomized into SHIPSS will be randomized into the Treatment Group and will receive hydrocortisone sodium succinate according to a predetermined dosing schedule.
  Interventions: Drug: Hydrocortisone, sodium succinate
- Placebo (Placebo Comparator): Approximately half of the subjects randomized into SHIPSS will be randomized into the Placebo Group and will receive equivalent study drug volumes of normal saline.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Hydrocortisone, sodium succinate — Patients randomized to the hydrocortisone treatment arm will receive an initial bolus of 2 mg/kg IV hydrocortisone, followed by 1 mg/kg (maximum 50 mg) of hydrocortisone dosed every six hours for a maximum of seven days or until all vasoactive infusions have been discontinued for at least 12 hours, whichever comes first. When the hydrocortisone course is completed, the medication will be discontinued.
  Other Names: SOLU-CORTEF- hydrocortisone sodium succinate injection
  Arms: Treatment
Drug: Normal saline — Patients randomized to the placebo treatment arm will receive an equivalent volume of normal saline, with the identical dosing schedule to the intervention (hydrocortisone) arm.
  Arms: Placebo

SUMMARY:
SHIPSS is a multi-institutional, prospective, controlled, randomized, double-blinded interventional trial that will examine the potential benefits and risks of adjunctive hydrocortisone prescribed for children with fluid and vasoactive-inotropic refractory septic shock.

It is hypothesized that adjunctive hydrocortisone will significantly reduce the incidence of new and progressive organ dysfunction (primary outcome) and proportion of children with poor outcomes, defined as death or severely impaired health-related quality of life (HRQL) (secondary outcome), as assessed at 28 days following study enrollment (randomization).

DETAILED DESCRIPTION:
Sepsis represents the most common cause of childhood mortality worldwide. In the United States alone, 200 cases of pediatric sepsis are diagnosed each day, with an associated hospital mortality rate of 5-10% and health care expenditures now approaching $5 billion annually. Moreover, nearly one third of children admitted to pediatric intensive care units (PICUs) for septic shock have not regained their baseline health-related quality of life one year following the sepsis event.

During early resuscitation of the child with septic shock, in addition to antibiotics, volume replacement, and vasoactive-inotropic support, the most recent pediatric treatment guidelines advise the practitioner to consider adjunctive hydrocortisone therapy if the patient "is at risk of absolute adrenal insufficiency or adrenal pituitary axis failure". However, the potential benefits and risks of this recommendation have not been rigorously examined. On the one hand, corticosteroids are inexpensive and have been frequently demonstrated to improve hemodynamic status in children and adults with sepsis. Conversely, this drug class is known to alter transcription of approximately 30% of the human genome. Notably, corticosteroids down regulate most aspects of the immune response, but particularly adaptive immunity. Moreover, recent data suggests that children with particular gene expression profiles in sepsis have increased likelihood of mortality when treated with corticosteroids.

SHIPSS (Stress Hydrocortisone In Pediatric Septic Shock) is a prospective, randomized, double-blinded, placebo-controlled trial examining the potential benefits and risks of adjunctive hydrocortisone prescribed to critically ill children with fluid and vasoactive-inotropic refractory septic shock. Up to 500 children will be enrolled, randomized, and evaluated at baseline, and 28 and 90 days following study enrollment.

The primary hypothesis is that hydrocortisone, compared to placebo, will decrease the the incidence of new or progressive organ dysfunction (primary outcome) and the proportion of subjects with poor outcomes, defined as death or severely impaired (≥25% decrease from baseline) HRQL (secondary outcome). Subjects will be monitored daily while receiving care in the PICU for the occurrence of adverse events, including the following protocol specified events:hyperglycemia treated with any insulin; gastrointestinal hemorrhage treated with blood product transfusion or vasopressin or octreotide infusion; delirium requiring medical treatment; and hospital-acquired infection treated with new antimicrobials. Finally, the investigators will test the hypothesis that biomarker-based prognostic and predictive enrichment strategies can improve our ability to identify which children with septic shock are more likely to benefit from adjunctive hydrocortisone, and which may be harmed. This trial will have a significant impact on public health by providing the heretofore missing evidence to inform guidelines regarding therapy for septic shock in children.

The SHIPSS trial will enroll patients from PICUs in Canada, the United States, Saudi Arabia, Israel, Brazil, Vietnam, Pakistan, Japan, Malaysia, and Singapore. Health Canada approval is not required as hydrocortisone is approved for use in septic shock in children, and this trial meets the criteria of a Phase IV study. In the United States, this trial is considered a Phase III trial as hydrocortisone is not approved for use in pediatric septic shock.

ELIGIBILITY:
Inclusion Criteria:

A child receiving treatment in a pediatric intensive care unit is eligible for recruitment into SHIPSS if she/he meets all of the following inclusion criteria:

1. Age is at least 1 month (with corrected gestational age ≥42 weeks), but less than 17 years and 8 months of age
2. A documented focus of infection or a strong suspicion of infection at PICU admission, or for patients who develop septic shock during PICU stay, at the onset of the septic shock event
3. Surveillance cultures (e.g. blood, urine, cerebral spinal fluid, wound) and/or other microbial diagnostic tests have been obtained
4. One or more antimicrobials have been prescribed
5. Core temperature >38.5 C or <36.0 C or leukocytosis or leukopenia (as defined by the local laboratory) or a left-shifted leukocyte differential (>10% immature granulocyte forms) or a neutrophil count of <0.5 x 109 cells per litre documented at least once within the 24 hours preceding screening
6. Treatment with a continuous infusion of vasoactive-inotropic agent(s) to maintain mean or systolic arterial blood pressure above the age-appropriate target set by the treating clinician
7. Administration of two or more vasoactive-inotropic agents at any dose or epinephrine or norepinephrine infusion(s) alone at greater than or equal to 0.10 mcg/kg/min for >1 hour.

Exclusion Criteria:

A child receiving treatment in a pediatric intensive care unit for sepsis is ineligible for enrollment into SHIPSS if she/he meets any of the following exclusion criteria:

1. All inclusion criteria have been present for > 12 hours
2. Attending physician expects to prescribe systemic corticosteroids for an indication other than septic shock
3. Patient has received any doses of systemic corticosteroids during treatment for sepsis
4. Enrolled concurrently in a competing interventional clinical trial (formal assessment to be conducted by SHIPSS Core Committee for each potential competing trial)
5. Etomidate or ketoconazole treatment within past 48 hours
6. Patient in whom steroids are contraindicated at time of screening (e.g. treatment for systemic fungal infection, cerebral malaria, strongyloides)
7. Known or suspected hypothalamic, pituitary or adrenal disease (including patient has received acute or chronic corticosteroid administration and the physician intends to provide corticosteroid for suspected adrenal suppression)
8. Attending physician, PICU care team, or legally recognized guardians not committed to full treatment and resuscitation at the time of screening
9. Patient documented to be pregnant
10. Previous enrollment in the SHIPSS study
11. Patient admitted directly to the PICU with a thermal burn who has been in the PICU for <72 hours prior to meeting SHIPSS inclusion criteria.
12. (U.S. sites only) Patient in the custody of US protective services
13. Patient being evaluated for brain death
14. Vasoactive-inotropic agents prescribed solely for an indication other than septic shock
15. Confirmed dengue fever

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2019-03-11 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
New or progressive multiple organ dysfunction syndrome as assessed utilizing the Pediatric Logistic Organ Dysfunction (PELOD-2) instrument. | 28 days following study enrollment
  Appearance of new or progression of existing organ dysfunctions according to PELOD-2 definitions. PELOD-2 considers 5 organ dysfunctions (neurological, cardiovascular, renal, respiratory, and hematological) with 10 total variables, with dysfunction scored 0 up to 6 for each organ category. Total minimum/maximal scores are 0/33, with increasing score indicating increasing risk of mortality. Logit (mortality) = -6.61 + 0.47 × PELOD-2 score. Probability of death = 1/(1 + exp [-logit(mortality)]). A new organ dysfunction or progression of organ dysfunction is defined as an increase score in any organ category from baseline.

SECONDARY OUTCOMES:
28-day hospital mortality or ≥25% decrease from baseline in health-related quality of life (HRQL) assessed utilizing the Pediatric Quality of Life Inventory, (PedsQL) | 28 days following study enrollment
  Mortality or ≥25% decrease in PedsQL from baseline

OTHER OUTCOMES:
SHIPSS specified adverse events | 28 days following study enrollment
  Occurrence of adverse events plausibly associated with corticosteroid administration. SHIPSS specified events include hyperglycemia, gastrointestinal hemorrhage, delirium, and hospital-acquired infection
Risk stratification sepsis biomarkers and pediatric sepsis endotype | Enrollment and Day 2
  Risk stratification sepsis biomarkers will be measured in serum obtained at enrollment and on Day 2. The PERSEVERE (PEdiatRic SEpsis biomarkEr Risk modEl) will be used to determine the patient's risk of mortality. mRNA will be isolated from blood samples collected at enrollment and on Day 2 to classify the patient as pediatric septic shock Endotype B or A. A composite outcome of sepsis endotype and PERSEVERE risk of mortality will be used to determine if a biomarker-based prognostic model and predictive enrichment strategies allow identification of children with septic shock more likely to benefit from adjunctive hydrocortisone. We hypothesize that pediatric septic shock "endotype B" subjects having an intermediate to high Pediatric Sepsis Biomarker Risk Model (PERSEVERE)-based risk of mortality will derive significant benefit from adjunctive corticosteroids, compared to endotype B subjects having a low risk and endotype A subjects at all risk levels.
Trichotomous mortality/morbidity outcome | 28 and 90 days following study enrollment
  This is a 3-level ordinal endpoint, with levels death, survival with severely impaired HRQL (≥25% decrease from baseline), and survival without severely impaired HRQL, assessed at 28 and 90 days. This approach is similar to that recently reported for assessment of functional status among children encountering critical illness, utilizing the Functional Status Scale. This endpoint is expected to be highly correlated with the primary efficacy endpoint.
90-Day Death or ≥25% decrease in HRQL from baseline | 90 days following study enrollment
  Mortality or ≥25% decrease in PedsQL from baseline
Vasoactive-inotropic infusion-free days through day 28 | 28 days following study enrollment
  Vasoactive-inotropic infusion-free days through day 28 is defined as 28 minus duration of vasoactive-inotropic infusions. Subjects who die or are still receiving vasoactive-inotropic infusions by day 28 will be censored at 28 days and assigned zero vasoactive-inotropic infusion-free days.
Mechanical ventilation-free days through day 28 | 28 days following study enrollment
  Mechanical ventilation-free days through day 28 is defined as 28 minus duration of mechanical ventilation. Subjects who die, are still receiving mechanical ventilation, or are transferred from the PICU still receiving mechanical ventilation by day 28 will be censored at 28 days and assigned zero mechanical ventilation-free days.
Utilization of acute renal replacement therapy (RRT) | Enrollment to PICU discharge, an average of 2 weeks
  Proportion of subjects receiving acute RRT. All types of acute RRT will be considered, including hemodialysis, continuous venovenous hemofiltration (CVVH), continuous venovenous hemodialysis (CVVHD), and peritoneal dialysis. RRT in patients on chronic RRT will not be considered.
Utilization of extracorporeal membrane oxygenation (ECMO) | Enrollment to PICU discharge, an average of 2 weeks
  Proportion of subjects receiving ECMO
Functional status - POPC | 28 and 90 days following study enrollment
  Gross functional status category staging will be made using the Pediatric Overall Performance Category (POPC) score.
Functional status - FSS | 28 and 90 days following study enrollment
  Functional Status Scale (FSS) will be employed to provide a more granular determination of changes in functional status.
PICU-free days through day 28 | 28 days following study enrollment
  PICU-free days through day 28 is defined as 28 minus duration of PICU stay. Subjects who die or are still in the PICU by day 28 will be censored at 28 days and assigned zero PICU-free days.
Hospital-free days through day 28 | 28 days following study enrollment
  Hospital-free days through day 28 is defined as 28 minus duration of hospital stay. Subjects who die or are still in the hospital by day 28 will be censored at 28 days and assigned zero hospital-free days through day 28.
Hospital-free days through day 90 | 90 days following study enrollment
  Hospital-free days through day 90 is defined as 90 minus duration of hospital stay. Subjects who die or are still in the hospital by day 90 will be censored at 90 days and assigned zero hospital-free days through day 90.
Need for new medical devices at hospital discharge | At time of hospital discharge, expected to be an average of 21 days from time of enrollment
  New medical devices prescribed at hospital discharge will be collected from the hospital discharge summary.
Frequency of primary care, specialty care, and emergency department visits and hospital readmissions | 90 days following study enrollment
  Enumeration of additional health care evaluations following the index hospital admission will occur by telephone survey at 90 days.
Disruption of family dynamics | Enrollment and 90 days following study enrollment
  The PedsQLTM 2.0 Family Impact Module will be used to quantify the impact of septic shock on family dynamics.
Cost Analysis - Cost of PICU admission for septic shock | 90 days following study enrollment
  The cost of each patients PICU admission will be determined by summing the cost of the following: PICU and hospital length of stay, frequency of primary care, specialty care, emergency department visits, and hospital readmissions up to 90 days following hospital discharge, new medical devices post hospital discharge and hospital costs of the admission for septic shock.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry J Zimmerman MD, MD, PhD, Principal Investigator — Seattle Children's Hospital, University of Washington School of Medicine; Michael Agus, MD, Principal Investigator — Boston Children's Hospital, Harvard Medical School; Mihir R Atreya, MD, MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati; David Wypij, PhD, Principal Investigator — Boston Children's Hospital, Harvard Medical School; Kusum Menon, MD, MSc, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (44):
- United States (18):
  - University of Arizona Medical Centre, Tucson, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital - Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Benioff Children's Hospital - San Francisco, San Francisco, California
  - Nemours Children's Health, Wilmington, Delaware
  - University of Chicago, Comer Children's Hospital, Chicago, Illinois
  - The University of Illinois at Chicago/OSF Children's Hospital of Illinois, Peoria, Illinois
  - University of Louisville, Norton Children's Hospital, Louisville, Kentucky
  - Boston Children's Hospital, Boston, Massachusetts
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital at Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Children's Hospital, Hershey, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin Health/American Family Children's Hospital, Madison, Wisconsin
- Brazil (2):
  - Santa Casa de Misericordia Da Bahia, Bahia
  - Hospital Jutta Batista - Rio de Janeiro, Rio de Janeiro
- Canada (10):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Centre hospitalier universitaire Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - Centre hospitalier de l'Université Laval, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Hadassah University Medical Center, Ein Kerem, Jerusalem
  - Schneider Children's Medical Center of Israel, Petah Tikva
- Japan (2):
  - Kobe Children's Hospital, Kobe
  - Aichi Children's Health and Medical Center, Nagoya
- Malaysia (3):
  - UKM Specialist Children's Hospital, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Sarawak General Hospital, Kuching
- Pakistan (2):
  - Shifa International Hospital, Islamabad
  - Aga Khan University Hospital, Karachi
- King Abdullah Specialist Children's Hospital, Riyadh, Saudi Arabia
- KK Women's and Children's Hospital, Singapore, Singapore
- Vietnam (2):
  - Vietnam National Children's Hospital, Hanoi
  - City Children's Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Per NIH policy, the SHIPSS investigators will provide a de-identified dataset and all the data-related documentation necessary to utilize the study data (dictionary, calculated variables, and standard operating procedures) to the NIH no later than 3 years after the final 90-day assessment or 2 years after the primary paper has been published, whichever comes first. The investigators will submit this dataset to the NICHD data repository, Data and Specimen Hub (DASH). In addition, final datasets and statistical analyses will be archived.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: No later than 3 years after the final 90-day assessment or 2 years after the primary paper has been published, whichever comes first.
Access Criteria: Anyone can access NICHD DASH, which is a public website with free access to the scientific research community. All users may browse and view information about studies and data archived in NICHD DASH. Users who are interested in submitting or requesting study data must register for a free account.

REFERENCES:
- [Derived] Menon K, Agus MSD, O'Hearn K, Coughlin-Wells K, Choong K, Kazzaz Y, Lee JH, McNally D, Atreya MR, Ramsay T, Watson RS, Wypij D, Zimmerman JJ; Stress Hydrocortisone in Pediatric Septic Shock (SHIPSS) Study Investigators, Canadian Critical Care Trials Group, and the Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Stress Hydrocortisone in Pediatric Septic Shock: Protocol for a Pragmatic, Multicenter, International, Randomized, Double-Blinded, Placebo-Controlled Interventional Trial. Pediatr Crit Care Med. 2026 Jan 1;27(1):102-113. doi: 10.1097/PCC.0000000000003872. Epub 2025 Nov 26. PMID 41504575
- [Derived] Tasker RC. Pediatric Critical Care Medicine: New Directions for 2026, Volume 27. Pediatr Crit Care Med. 2026 Jan 1;27(1):1-2. doi: 10.1097/PCC.0000000000003874. Epub 2026 Jan 8. No abstract available. PMID 41504572
- [Derived] Basu S, Habet V, Delgado M, Chiu P, Knox D, Thibault E, Shukla A, Harrington E, Bailey V, Lipsitz S, Fu Y, Agus M, Kheir J, Sasaki J, Moynihan K. Adjunctive Corticosteroids for Hypotension in the Pediatric Cardiac ICU: Single-Center Retrospective Study, 2020-2021. Pediatr Crit Care Med. 2025 Jul 1;26(7):e877-e888. doi: 10.1097/PCC.0000000000003757. Epub 2025 May 1. PMID 40310269
- See also: Website for SHIPSS investigation — http://www.shipss.org